CLINICAL TRIAL: NCT05092945
Title: Quantifying Brown Adipose Tissue Thermogenesis in Type 2 Diabetes
Brief Title: Brown Adipose Tissue Metabolism in Type 2 Diabetes
Acronym: GB8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, André Carpentier, tenured professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-2990
Record Dates: First submitted 2021-05-19; First posted 2021-10-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Niacin

STUDY DESIGN:
Intervention Model Description: Two groups in parallel (with and without Type 2 diabetes). In each group, the protocol will be carried out as a within-subject, randomized, cross-over study in which each subject will serve as his/her own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Subject with Type 2 Diabetes- cold exposure (Active Comparator): 3-hour cold exposure: Protocol B
  Interventions: Other: Cold exposure
- Subject with type 2 Diabetes- cold exposure and nicotinic acid (Experimental): 3-hour cold exposure with oral nicotinic acid: Protocol A
  Interventions: Other: Cold exposure; Drug: Oral Nicotinic acid
- Subject without Type 2 Diabetes- cold exposure (Active Comparator): 3-hour cold exposure: Protocol B
  Interventions: Other: Cold exposure
- Subject without type 2 Diabetes- cold exposure and nicotinic acid (Experimental): 3-hour cold exposure with oral nicotinic acid: Protocol A
  Interventions: Other: Cold exposure; Drug: Oral Nicotinic acid

INTERVENTIONS:
Other: Cold exposure — The liquid-conditioned tube suit will be perfused with 18°C water using a temperature- and flow-controlled circulation bath from time 0 to 180 min.
Drug: Oral Nicotinic acid — A total of 500 mg of nicotinic acid will be given orally, at a rate of 2 doses of 150 mg and 2 doses of 100 mg: one dose of 150 mg at time 0 and 60 minutes, one dose of 100 mg at time 120 minutes and 180 minutes.
  Other Names: Niacin 500 (Jamp Pharma) NPN 00557412
  Arms: Subject with type 2 Diabetes- cold exposure and nicotinic acid; Subject without type 2 Diabetes- cold exposure and nicotinic acid

SUMMARY:
Activation of brown adipose tissue (BAT) by cold exposure.

BAT thermogenesis and BAT volume of metabolic activity will be assessed by Positron-Emitting-Tomography (PET/CT) and MRI/MRS imaging and new pharmacological methods to modulate BAT thermogenesis.

All previous data on the functioning of Brown Adipose Tissue (BAT) were obtained by Positron-Emitting-Tomography (PET) imaging studies using fluorodeoxyglucose F18 ( [18F]- FDG). This approach underestimates the actual activity of the BAT. In this study, the investigator is going to use a new PET tracer (C11-palmitate) which is a fat molecule. This will allow to quantify more accurately the activity of brown fat.

DETAILED DESCRIPTION:
The study protocol includes three visits: the screening visit (V1) and two PET/MRI imaging studies (V2 and V3) performed in random order at an interval of 7 to 14 days.

PET/ MRI studies will be performed with and without nicotinic acid. A total of 500 mg of nicotinic acid will be given orally, at a rate of 2 doses of 150 mg and 2 doses of 100 mg, through V2 (protocol A): one dose at time 0, 60 minutes, 120 minutes and 180 minutes.

During V2 and V3, participants will undergo Acute Cold Exposure to stimulate brown adipose tissue.

The morning of each PET imaging study, the participants will follow an MRI acquisition to determine hepatic, pancreatic, visceral and BAT lipid content, followed by an MRS acquisition in the hepatic and cervico-thoracic region. MRI and MRS acquisition of the hepatic and cervico-thoracic region will be repeated again at the end of the day.

The radioactive PET tracers used in this study are the [11C]-acetate, [11C]-palmitate and [18F]-FDG followed by dynamic and whole-body scans.

Stable isotopes such as [U-13C]-palmitate (0.08 umol/kg/min), 5D-glycérol (0.1 µmol/kg/min,) and tritiated glucose (of 1.5 uCi/min) will be perfused from the start of the day until time 180 min.

ELIGIBILITY:
Inclusion Criteria:

* 10 men and 10 women with T2D.
* 10 non-diabetic men and 10 non-diabetic women (matched for sex, BMI and age to the T2D participants).

Exclusion Criteria:

* Change in weight of more than 2 kg over the past 3 months or recent changes in lifestyle;
* Treatment with a fibrate, thiazolidinedione, insulin, beta-blocker, GLP-1 agonist, or other drug known to affect lipid or carbohydrate metabolism, except statins, metformin, sulfonylurea, DPP-IV inhibitor and other antihypertensive agents that can be temporarily stopped safely prior to the studies, as per our approved protocols;
* Presence of overt cardiovascular, liver, renal or other medical conditions;
* Smoking or consumption of more than 2 alcoholic beverages per day;
* Any other contraindication to temporarily suspending current medications for lipids or hypertension;
* Any contraindication to MRI scanning.
* Having participated to a research study with exposure to radiation in the last two years before the start of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
BAT volume | 180 minutes after the start of the cold exposure
  Assessed using i.v. injection of 18FDG with whole-body PET/CT acquisition.
Brown Adipose Tissue (BAT) Glucose uptake | 150 minutes after the start of the cold exposure
  Assessed using i.v. injection of 18FDG with sequential dynamic PET/CT scanning

SECONDARY OUTCOMES:
Activation of BAT (oxidative metabolism) | 90 minutes after beginning cold exposure
  Measured with 11C-acetate using dynamic PET/CT acquisition.
Fatty Acid uptake and metabolism | at baseline and at time 120 minutes after beginning cold exposure
  Measured with 11C-palmitate using dynamic PET/CT acquisition.
BAT triglyceride content | at baseline and at time 180 (for CT) and 240 (for MR) after cold exposure.
  Estimated by CT and MR using 1H-MRS and Dixon sequences on a 3T clinical MRI system.
Whole-body lipolysis | -150 and 0 minutes before and 60, 120 and 180 minutes after cold exposure.
  Systemic appearance rate of glycerol and fatty acid determined by perfusion of [1,1,2,3,3-2H]-glycerol, [U-13C]-palmitate tracers and concentration of total NEFA, triglycerides, palmitate, oleate, linoleate, glycerol.
Hepatic Glucose production | -150 and 0 minutes before and 60, 120 and 180 minutes after cold exposure.
  Systemic appearance rate of glucose determined by perfusion of [3-3H]-glucose.
Substrate utilisation | -150 and 0 minutes before and 60, 120 and 180 minutes after cold exposure.
  VO2 and VCO2 will be measured by indirect calorimetry to calculate carbohydrate and fatty acid oxidation rates.
Changes in insulin level and secretion | -150 and 0 minutes before and 60, 120 and 180 minutes after cold exposure.
  measured with ELISA and Milliplex.

CONTACTS AND LOCATIONS:
Overall Officials: André Carpentier, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS, Sherbrooke, Quebec, Canada